CLINICAL TRIAL: NCT03976479
Title: Body Composition, Nutritional and Cardiovascular Status and Lifestyle Factors of Adults Who Are on Short-, Medium- and Long-term Plant-Based Diet
Brief Title: Body Composition, Nutritional and Cardiovascular Status and Lifestyle Factors of Adults Who Are on Plant-Based Diet
Acronym: SuppWFPBD
Status: Completed | Type: Observational
Sponsor: Boštjan Jakše (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor-Investigator, Boštjan Jakše, Physical education teacher (Phd student of Nutrition), Barbara Jakše s.p.
Organization: Barbara Jakše s.p. (Other)
Other Study IDs: KR3
Record Dates: First submitted 2019-06-01; First posted 2019-06-06 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Conditions Influencing Health Status; Body Weight; Lipid Metabolism Disorders; Uricemia; Blood Pressure Disorders; Physical Stress; Sleep Disorder; Stress, Psychological
Keywords: Body composition; Nutritional status; Lipids; Blood pressure; Lifestyle factors
MeSH Terms: conditions — Body Weight; Lipid Metabolism Disorders; Hyperuricemia; Sleep Wake Disorders; Stress, Psychological | interventions — Body Composition; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Body composition, questionnaires, biochemistry and blood pressure results — Body composition status, nutritional status, cardiovasculat status, health status, lifestyle factors

SUMMARY:
There is an objective lack of data on the body composition, nutritional status, cardiovascular status and lifestyle of adults on a plant-based diet (PBD). The aim in this cross-sectional study investigators will document the differences in the body composition, nutritional intake and general health status of healthy adults aged 18 to 80 years who are on plant-based diet of 0.5-10 years and to determine if their body composition status is associated to the duration of eating with PBD between the 3 groups: those that are 0.5-2 years (short-term), 2-5 years (medium-term) and 5-10 years (long-term) on PBD.

This study will also include the monitoring of other factors of healthy and active lifestyle of PBD participants, namely the status of habitual and organized physical activity, the status of daily long-term seating, the status of stress and hygiene of sleep, socio-economic status and the motive(s)/reasons for starting PBD. Investigators will also record their maximum (lifetime) body weight, body weight upon entering the PBD lifestyle, and using data from participants, blood analysis to collect their basic biochemistry results, and data on current blood pressure status.

The investigators hypothesis is that:

(H1): There are no differences in nutritional status between people who are short- (0.5-2 years), the medium- (2-5 years) or the long-term (5-10 years) on PBD.

(H2): At least 80% of the tested subjects have plasma lipid values and blood pressure within the reference values.

(H3): There is difference in lipid profile and body composition between people who are short- and the medium but not between medium and long-term PBD.

DETAILED DESCRIPTION:
In the study investigators will voluntarily enroll all participants within inclusion/exclusion criteria that are willing to participate in the study. Investigators will anticipate that for approx. 150-200 healthy adult PBD participants investigators will require approx. 2555 invited and interviewed candidates, of both sexes, aged 18-80 years, without restrictions on current body mass index (BMI) status, that are on PBD for 0.5-10 years and live a healthy and active lifestyle.

The methods to be used are a medically approved bioimpedance body composition monitor (Tanita, 780 S MA, Tokyo, Japan), medically approved body weight scale and body height gauge (MPE 250K100HM), a 3-day dietary record (3-DR), one adopted by NIH: socio-demographic, economic status and motive for PBD questionnaire, and three standardized questionnaires: (1) habitual and organized physical activity, and the frequency of sitting (IPAQ-long), (2) stress (PSQ-30), and (3) quality of sleep (PSQI).

Concerning 3-DR, the study participants will weight and record all foods, beverages consumed, as well as leftovers, and dietary supplements over three consecutive days (two weekdays and one weekend) using electronic kitchen scales. The study participants will choose the day of the beginning of dietary recording within a given period (i. e.: Sunday, Monday, Tuesday or Thursday, Friday, Saturday). When exact weighing will not be possible (e.g., in case of eating out), household measures (spoon, cup, glass, etc.) and a picture book with household measures in adults' portion sizes (photos of reference foods with their actual gram weight) (NIJZ, 2016), allowed semi-quantitative recording. For the evaluation of dietary intake, investigators will use dietary software, Open Platform for Clinical Nutrition (OPEN), which is a web-based application (http://opkp.si/) and has been developed by the Jozef Stefan Institute and supported by the EuroFIR AISBL (http://eurofir.org) and the European Federation of the Association of Dietitians (EFAD). Dietary software has been upgraded to 3-DR methodology.

Food intake data (from 3-DR) will be used for assessment of energy, macro- and micronutrients intakes using OPEN. The energy and nutrient contents of commercial food or home prepared foods, will estimated by recipe simulation using labelled ingredients and nutrient contents. OPEN will be continuously updated by adding those products or recopies recorded by study participants on PBD.

In order to assess the nutritional intake from dietary supplements, we will use Res-Pons d.o.o. services, which professionally manages the database with all dietary supplements products on the Slovenian market (Pretehtajte.si, 2018).

Investigators will also record their maximum (lifetime) body weight, body weight upon entering the PBD lifestyle, and using data taken blood analysis to collect their basic biochemistry results, measured in a standard and comparable method (plasma lipids, uric acid and a hemogram), and data on current blood pressure status.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age from 18-80 years, on PBD longer than 0.5 years.
* PB dieters who may have some kind of food intolerance or food restriction (e.g. gluten, tomato, peanuts, citrus, etc.).
* No restriction on participants current BMI
* Knowing (BIA measured) PB dieters baseline BM and fat %
* Currently smoking tobacco products is not an exclusion criterion, but we will record it and report in demographic data

Exclusion Criteria:

* Adults on PBD but with active diseases (e.g. cardiovascular diseases, type 2 diabetes, cancer, autoimmune and neurodegenerative disease ect.).
* Adults on PBD with the current use of drugs for measured blood markers (lipids and blood pressure).
* Without major musculoskeletal restrictions
* Pregnant and lactating woman
* Currently competitive or top level athletes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heatlhy and active long-term PB dieters
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Body weight status | Cross-sectional (June-July 2019)
  Body weight measured with medically approved weighing scale
Height status | Cross-sectional (June-July 2019)
  Height status measured with medically approved weighing scale with height rod
Body mass index (BMI) status | Cross-sectional (June-July 2019)
  Measured weight and height will be combined to report BMI in kg/m^2
Lean tissue mass status | Cross-sectional (June-July 2019)
  Lean tissue mass measured with medically approved bioimpedance analysis
Fat tissue mass status | Cross-sectional (June-July 2019)
  Fat tissue mass measured with medically approved bioimpedance analysis
Nutritional status | Cross-sectional (June-July 2019)
  Nutrititional status measured with 3-day dietary record (3-DR)
Serum cholesterol status | Cross-sectional (June-July 2019)
  Serum total cholesterol concentration
Oxidized Low Density Lipoprotein (LDL)-cholesterol status | Cross-sectional (June-July 2019)
  Serum concentration of oxidized LDL-cholesterol
Serum HDL cholesterol status | Cross-sectional (June-July 2019)
  Serum HDL cholesterol contentration
Serum triglyceride status | Cross-sectional (June-July 2019)
  Serum triglyceride concentrations
Blood pressure status | Cross-sectional (June-July 2019)
  Blood pressure status

SECONDARY OUTCOMES:
Socio-economic and demographic status | Cross-sectional (June-July 2019)
  Socio-economic and demographic status measured using Nutritional behaviours of adults Slovenians from the point of of health prevention questionnaire (Slovenian NIH)
Physical activity status | Cross-sectional (June-July 2019)
  Physical activity status measured by The International Physical Activity Questionnaires (IPAQ)
Stress status | Cross-sectional (June-July 2019)
  Stress status measured with Perceived Stress Questionnaire (PSQ)
Sleep status | Cross-sectional (June-July 2019)
  Sleep status measured with The Pittsburgh Sleep Quality Index (PSQI)
Serum uric acid status | Cross-sectional (June-July 2019)
  Serum uric acid concentration (safety outcome)
Hemoglobin status | Cross-sectional (June-July 2019)
  Hemoglobin concentration (safety outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- PDP Spodnje Črnuče, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karlsen MC, Rogers G, Miki A, Lichtenstein AH, Folta SC, Economos CD, Jacques PF, Livingston KA, McKeown NM. Theoretical Food and Nutrient Composition of Whole-Food Plant-Based and Vegan Diets Compared to Current Dietary Recommendations. Nutrients. 2019 Mar 14;11(3):625. doi: 10.3390/nu11030625. PMID 30875784
- [Background] Melina V, Craig W, Levin S. Position of the Academy of Nutrition and Dietetics: Vegetarian Diets. J Acad Nutr Diet. 2016 Dec;116(12):1970-1980. doi: 10.1016/j.jand.2016.09.025. PMID 27886704
- [Background] Satija A, Bhupathiraju SN, Spiegelman D, Chiuve SE, Manson JE, Willett W, Rexrode KM, Rimm EB, Hu FB. Healthful and Unhealthful Plant-Based Diets and the Risk of Coronary Heart Disease in U.S. Adults. J Am Coll Cardiol. 2017 Jul 25;70(4):411-422. doi: 10.1016/j.jacc.2017.05.047. PMID 28728684
- [Background] Willett W, Rockstrom J, Loken B, Springmann M, Lang T, Vermeulen S, Garnett T, Tilman D, DeClerck F, Wood A, Jonell M, Clark M, Gordon LJ, Fanzo J, Hawkes C, Zurayk R, Rivera JA, De Vries W, Majele Sibanda L, Afshin A, Chaudhary A, Herrero M, Agustina R, Branca F, Lartey A, Fan S, Crona B, Fox E, Bignet V, Troell M, Lindahl T, Singh S, Cornell SE, Srinath Reddy K, Narain S, Nishtar S, Murray CJL. Food in the Anthropocene: the EAT-Lancet Commission on healthy diets from sustainable food systems. Lancet. 2019 Feb 2;393(10170):447-492. doi: 10.1016/S0140-6736(18)31788-4. Epub 2019 Jan 16. No abstract available. PMID 30660336
- See also: NIJZ, Slikovno-gradivo-za-dolocanje-vnosa-zivil, 2016. Available at: http://www.nijz.si/sl/publikacije/slikovno-gradivo-za-dolocanje-vnosa-zivil , assesed 30.05.2019 — http://www.nijz.si/sl/publikacije/slikovno-gradivo-za-dolocanje-vnosa-zivil
- See also: OPEN Platform for Clinical Nutrition — http://opkp.si/
- See also: EuroFIR AISBL — http://eurofir.org
- See also: Res Pons d.o.o. — https://pretehtajte.si/